CLINICAL TRIAL: NCT03724942
Title: A Multicenter, Uncontrolled, Open-label Trial to Evaluate the Safety of Extended Treatment With Brexpiprazole (OPC-34712) to Patients With Agitation Associated With Dementia of the Alzheimer's Type
Brief Title: Brexpiprazole for the Long-term Treatment of Patients With Agitation Associated With Dementia of the Alzheimer's Type
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 331-102-00184; JapicCTI-184179 (Other: Japic)
Record Dates: First submitted 2018-10-28; First posted 2018-10-30 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Agitation Associated With Dementia of the Alzheimer's Type
MeSH Terms: interventions — brexpiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brexpiprazole (Experimental)
  Interventions: Drug: Brexpiprazole

INTERVENTIONS:
Drug: Brexpiprazole — Brexpiprazole 1mg or 2mg will be orally once daily for 14 weeks
  Other Names: OPC-34712

SUMMARY:
To evaluate the safety of brexpiprazole 1 mg or 2 mg after a 14 week treatment regimen for agitation associated with dementia of the Alzheimer's type patients who completed in a double-blind trial, and to investigate the efficacy of brexpiprazole.

ELIGIBILITY:
Inclusion Criteria:

* Patients who completed the double-blind treatment period for 10 weeks and all observation, examination and evaluation at Week 10 of the double-blind trial.
* Patients whose caregiver can properly collect the necessary information.

Exclusion Criteria:

* Patients who had a serious adverse event which the principal investigator or sub-investigator assessed as related to the investigator product during the double-blind trial.
* Patients who had delirium during the double-blind trial.

Ages: 55 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2022-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Osamu Sato, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Jisenkai Nanko Psychiatric Institute, Shirakawa, Japan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal.
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article Publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com.

REFERENCES:
- [Derived] Nakamura Y, Adachi J, Hirota N, Iba K, Shimizu K, Nakai M, Mori N, Takahashi K. Long-term safety and tolerability of brexpiprazole for Japanese patients with agitation in Alzheimer's disease dementia: A multicenter, open-label study. J Alzheimers Dis Rep. 2025 Apr 16;9:25424823251334054. doi: 10.1177/25424823251334054. eCollection 2025 Jan-Dec. PMID 40290781

RESULTS

PARTICIPANT FLOW:
Groups:
- ROLLOVER BREX: Rollover subjects from the brexpiprazole group in Trial 331-102-00088
- ROLLOVER PLACEBO: Rollover subjects from the placebo group in Trial 331-102-00088
Period: Overall Study
Arm/Group | ROLLOVER BREX | ROLLOVER PLACEBO
Started | 102 | 62
Completed | 73 | 44
Not Completed | 29 | 18
Not completed — Adverse Event | 20 | 14
Not completed — Lack of Efficacy | 0 | 1
Not completed — Physician Decision | 5 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Bedridden All Day and Required Full Assistance for Excretion, Meals and Change of Clothes | 0 | 1
Not completed — Withdrawal by Legal Representative | 3 | 0

BASELINE CHARACTERISTICS:
Population: This trial was conducted in 164 participants in Japan.
Groups:
- Total: Total of all reporting groups
Arm/Group | ROLLOVER BREX | ROLLOVER PLACEBO | Total
Number analyzed (Participants) | 102 | 62 | 164
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 2 | 8
  >=65 years | 96 | 60 | 156
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.0 (6.8) | 80.2 (6.9) | 79.5 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 36 | 101
  Male | 37 | 26 | 63
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 102 | 62 | 164
Region of Enrollment [Number; unit: participants]
  Japan | 102 | 62 | 164

OUTCOME MEASURES:

1. Primary Outcome: The Frequency of Subjects With Treatment-Emergent Adverse Events (TEAEs)
Description: This trial enrolled subjects rolled over from Trial 331-102-00088, and the safety of brexpiprazole when administered for a maximum of 24 weeks (including the treatment period of Trial 331-102-00088) was evaluated.
Time Frame: From baseline to week 14
Population: The safety analysis set comprised subjects who have received at least 1 dose of the IMP.
Measure: Number; unit: Percentage of percipitante
Arm/Group | ROLLOVER BREX | ROLLOVER PLACEBO
Number analyzed (Participants) | 102 | 62
Percentage of percipitante | 90.2 | 90.3

2. Secondary Outcome: Mean Change From Baseline in Cohen-Mansfield Agitation Inventory (CMAI) Score at 14 Weeks After Dosing
Description: The CMAI assessed the frequency of agitated behaviors in elderly persons, such as hitting, cursing, and restlessness. It consisted of 29 items all rated on a 1 to 7 scale with 1 being the "best" rating and 7 being the "worst" rating. The minimum possible CMAI total score was 29, and the maximum possible CMAI total score was 203. A decrease in score indicated improvement in symptoms.
Time Frame: Baseline and 14 weeks after dosing
Population: The efficacy analysis set will comprise subjects who have received at least 1 dose of the IMP and from whom CMAI total scores have been obtained at baseline and at least 1 time point after initiation of treatment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | ROLLOVER BREX | ROLLOVER PLACEBO
Number analyzed (Participants) | 96 | 60
Units on a scale | -2.5 (9.9) | -6.4 (9.3)

3. Secondary Outcome: Mean Change From Baseline in Clinical Global Impression of Severity (CGI-S) Score at 14 Weeks After Dosing.
Description: The CGI-S was used to rate the severity of agitation. Scores were: 0 = not assessed; 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill participants. A decrease in score indicated improvement in symptoms.
Time Frame: Baseline and 14 weeks after dosing.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | ROLLOVER BREX | ROLLOVER PLACEBO
Number analyzed (Participants) | 96 | 60
Units on a scale | -0.2 (0.8) | -0.4 (1.1)

4. Secondary Outcome: Clinical Global Impression of Improvement (CGI-I) Score at 14 Weeks After Dosing
Description: The CGI-I Scale was clinician-rated scale which assessed the total improvement of the patient's condition compared to that at baseline. Scores range from 0 to 7: 0 = Not assessed, 1= Very much improved, 2 = Much improved, 3= Minimally improved, 4= No change, 5= Minimally worse, 6= Much worse, 7= Very much worse. Higher scores indicate worse condition.
Time Frame: 14 weeks after dosing.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | ROLLOVER BREX | ROLLOVER PLACEBO
Number analyzed (Participants) | 96 | 60
Units on a scale | 3.1 (1.2) | 2.7 (1.1)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from signing of the informed consent form through 35 days after last dose of study drug (Up to approximately Week 19)
Description: Subjects who received at least one dose of IMP were included in the safety analysis.
Arm/Group | ROLLOVER BREX | ROLLOVER PLACEBO
All-Cause Mortality (participants affected / at risk) | 0/102 | 1/62
Serious Adverse Events (participants affected / at risk) | 7/102 | 4/62
Other Adverse Events (participants affected / at risk) | 90/102 | 55/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ROLLOVER BREX (N=102) | ROLLOVER PLACEBO (N=62)
Gait disturbance (General disorders) | 2 | 0
Pneumonia (Infections and infestations) | 1 | 1
Pneumonia aspiration (Infections and infestations) | 1 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 1 | 0
Akathisia (Nervous system disorders) | 1 | 0
Bradykinesia (Nervous system disorders) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ROLLOVER BREX (N=102) | ROLLOVER PLACEBO (N=62)
Dry eye (Eye disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 8 | 3
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Salivary hypersecretion (Gastrointestinal disorders) | 6 | 4
Vomiting (Gastrointestinal disorders) | 1 | 2
Gait disturbance (General disorders) | 5 | 3
Oedema (General disorders) | 1 | 3
Pyrexia (General disorders) | 4 | 4
Peripheral swelling (General disorders) | 1 | 3
Hepatic function abnormal (Hepatobiliary disorders) | 3 | 1
Conjunctivitis (Infections and infestations) | 2 | 2
Herpes zoster (Infections and infestations) | 1 | 2
Nasopharyngitis (Infections and infestations) | 5 | 4
Tinea pedis (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 3 | 2
Fall (Injury, poisoning and procedural complications) | 12 | 4
Femur fracture (Injury, poisoning and procedural complications) | 0 | 2
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 8 | 5
Wound (Injury, poisoning and procedural complications) | 3 | 4
Skin laceration (Injury, poisoning and procedural complications) | 0 | 3
Skin abrasion (Injury, poisoning and procedural complications) | 11 | 2
Blood albumin decreased (Investigations) | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 0 | 3
Weight decreased (Investigations) | 5 | 2
Weight increased (Investigations) | 1 | 2
Hepatic enzyme increased (Investigations) | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0
Decreased appetite (Metabolism and nutrition disorders) | 5 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 9 | 4
Akathisia (Nervous system disorders) | 4 | 2
Bradykinesia (Nervous system disorders) | 9 | 3
Dyskinesia (Nervous system disorders) | 3 | 1
Dystonia (Nervous system disorders) | 3 | 2
Extrapyramidal disorder (Nervous system disorders) | 3 | 6
Headache (Nervous system disorders) | 1 | 2
Parkinsonism (Nervous system disorders) | 4 | 3
Seizure (Nervous system disorders) | 0 | 2
Somnolence (Nervous system disorders) | 13 | 7
Tremor (Nervous system disorders) | 4 | 3
Sedation complication (Nervous system disorders) | 7 | 9
Insomnia (Psychiatric disorders) | 5 | 12
Restlessness (Psychiatric disorders) | 0 | 2
Urinary incontinence (Renal and urinary disorders) | 3 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 4 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 2
Skin exfoliation (Skin and subcutaneous tissue disorders) | 4 | 1
Internal haemorrhage (Vascular disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-02-03): https://cdn.clinicaltrials.gov/large-docs/42/NCT03724942/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-04): https://cdn.clinicaltrials.gov/large-docs/42/NCT03724942/SAP_001.pdf